CLINICAL TRIAL: NCT01776463
Title: A Single Centre, Randomized, Double-blind, Ascending Dose, Placebo-controlled, and Food Effect Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Doses of Z-360 and Placebo in Healthy Subjects
Brief Title: A Healthy Subject Study With Z-360 and Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01A10101
Record Dates: First submitted 2013-01-15; First posted 2013-01-28 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Healthy Volunteers
Keywords: Z-360; Japanese; pK
MeSH Terms: interventions — Z-360

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Z-360 (Experimental): 1)Single dose study (60, 120, 240, 480, 720mg), 2)Food effect study(120mg), 3)Multiple doses study(120, 240mg (BID))
  Interventions: Drug: Z-360
- Placebo (Placebo Comparator): 1)Single dose study, 2)Multiple doses study
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Z-360
  Arms: Z-360
Drug: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics (including food effect) of single and multiple doses of Z-360 in healthy Japanese subjects.

DETAILED DESCRIPTION:
This is a single centre, randomized, double-blind, placebo-controlled, parallel-group, and food effect study.This is three parts study. The purpose of the first part (Part 1) is the evaluation of the safety, tolerability, and pharmacokinetics after single ascending doses of Z-360.The second part (Part 2 ) is the evaluation of the pharmacokinetics of food effect of Z-360.The third part (Part 3) is the evaluation of the safety, tolerability, and pharmacokinetics after multiple ascending doses of Z-360.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between 20 to 49 years of age inclusive
2. Body mass index (BMI) within the range 17.6 to 26.4 kg/m2 inclusive
3. The subject is capable of giving written informed consent prior to admission into this study

Exclusion Criteria:

1. History or presence of drug hypersensitivity, drug dependence, narcotic dependence or alcohol dependence
2. History or presence disease of digestive, liver, kidney, blood, cardiovascular, neuropsychiatric which may affect participation or results of this study
3. Positive test for Hepatitis B surface antigen, Hepatitis C antibody, HIV antigen antibody or Serological test for syphilis
4. Use of any medication within 1 week prior to dosing
5. Received any investigational drugs with new active ingredients within 16 weeks prior to dosing the study or received any investigational drugs in other clinical studies within 12 weeks
6. Whole blood collection exceeding 200 mL within 4 weeks, apheresis within 2 weeks, or blood withdrawal exceeding 400 mL within 12 weeks (blood donation, etc) prior to dosing
7. Others, patients who are unfit for the study as determined by the attending physician

Ages: 20 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
General safety and tolerability endpoints: (Adverse events, Vital signs, 12-lead ECG and clinical laboratory safety tests) | up to 6 weeks

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of single and multiple doses of Z-360 in healthy subjects | up to 6 weeks
  pK (AUC, Cmax, Tmax, T1/2, MRT, CL/F, V/F)

CONTACTS AND LOCATIONS:
Overall Officials: Eri Sato, MD, Principal Investigator — Sumida
Locations (1):
- Sumida, Sumida-ku, Tokyo, Japan